CLINICAL TRIAL: NCT05092490
Title: Serratus Anterior Plane Block Combined With Transversus Thoracic Muscle Plane Block Versus Conventional Local Anesthetic Infiltration for SICD Implantation: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Joel Yarmush, Program Director, Department of Anesthesiology, Principal Investigator, Clinical Professor, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1723038-1
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Serratus Anterior Plane Block; Transversus Thoracis Plane Block; Subcutaneous ICD
Keywords: Serratus anterior plane block; Transversus thoracis plane block; SICD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not informed about which block they are receiving
  1 study personnel assess the pain scores and patient satisfaction postoperative
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined serratus anterior plane block and transversus thoracis plane block (Experimental): The study group will receive a combined plane block by a dedicated anesthesia team prior to their procedure. 20 mL of local anesthetic (0.25% bupivacaine) will be injected for the Serratus anterior plane block and another 20 mL of local anesthetic (0.25% bupivacaine) will be injected in transversus thoracis plane block
  Interventions: Procedure: Combined serratus anterior plane block and transversus thoracis plane block
- Stand local anesthetic infiltration (Active Comparator): Local anesthetic infiltration of the incision sites will be performed by the cardiologist prior to, and as, necessary during the procedure. The amount of local anesthetic used will be determined intraoperatively by the cardiologist according to the patients' requirements.
  Interventions: Procedure: Standard local infiltration technique

INTERVENTIONS:
Procedure: Combined serratus anterior plane block and transversus thoracis plane block — The study group will receive a combined plane block by a dedicated anesthesia team prior to their procedure. 20 mL of local anesthetic (0.25% bupivacaine) will be injected for the Serratus anterior plane block and another 20 mL of local anesthetic (0.25% bupivacaine) will be injected in transversus thoracis plane block
  Arms: Combined serratus anterior plane block and transversus thoracis plane block
Procedure: Standard local infiltration technique — Local anesthetic infiltration of the incision sites will be performed by the cardiologist prior to, and as, necessary during the procedure. The amount of local anesthetic used will be determined intraoperatively by the cardiologist according to the patients' requirements.
  Arms: Stand local anesthetic infiltration

SUMMARY:
This is a prospective randomized study. The aim is to investigate the efficacy of a combined SAPB with TTPB for perioperative pain control compared to the standard local anesthetic infiltration technique in adult patients undergoing SICD implantation. The hypothesis is that the combined plane block provides better pain control compared to the standard local infiltration technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to provide a written informed consent.
* Patient is scheduled to have an elective SICD implantation procedure.
* Patient has none of the exclusion criteria

Exclusion Criteria:

* Patient is unable to provide a written informed consent.
* Patient is younger than 18 years old.
* Patients with prior thoracotomy or other thoracic surgery altering anatomy.
* Patients with neurological deficits.
* Patients with impaired coagulation (Platelet count < 50,000 cells/mcl and/or INR > 1.4).
* Patient on anticoagulation therapy.
* Patient's weight below 50 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score measured | 1 day
  by Numerical Rating Scale pain (0-10), 0 is no pain, 10 is the worst

SECONDARY OUTCOMES:
Intraoperative pain score measured | Intraoperative
  by Numerical Rating Scale pain
Intraoperative sedation score | Intraoperative
  Richmond Agitation Sedation Scale (RASS) (+4 to -5) +4 combative
  -5 unarousable
Total local anesthetic volume used | Intraoperative
  Total local anesthetic volume used
Procedure duration | Intraoperative
  Procedure duration
Intraoperative hemodynamics | Intraoperative
  Intraoperative hemodynamics
Time to 1st rescue pain medication | 1 day
  Time to 1st rescue pain medication after surgery
Postoperative opioid consumption | 1 day
  Amount of opioids consumed after surgery
Patient satisfaction | 1 day
  How much is the patient satisfied with the pain management in the perioperative period
Block related complications | 1 day
  Any complications that may happen from either blocks, e.g infection, bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Result] Burke MC, Gold MR, Knight BP, Barr CS, Theuns DAMJ, Boersma LVA, Knops RE, Weiss R, Leon AR, Herre JM, Husby M, Stein KM, Lambiase PD. Safety and Efficacy of the Totally Subcutaneous Implantable Defibrillator: 2-Year Results From a Pooled Analysis of the IDE Study and EFFORTLESS Registry. J Am Coll Cardiol. 2015 Apr 28;65(16):1605-1615. doi: 10.1016/j.jacc.2015.02.047. PMID 25908064
- [Result] Weiss R, Knight BP, Gold MR, Leon AR, Herre JM, Hood M, Rashtian M, Kremers M, Crozier I, Lee KL, Smith W, Burke MC. Safety and efficacy of a totally subcutaneous implantable-cardioverter defibrillator. Circulation. 2013 Aug 27;128(9):944-53. doi: 10.1161/CIRCULATIONAHA.113.003042. PMID 23979626
- [Result] Essandoh MK, Otey AJ, Abdel-Rasoul M, Stein EJ, Turner KR, Joseph NC, Daoud EG. Monitored Anesthesia Care for Subcutaneous Cardioverter-Defibrillator Implantation: A Single-Center Experience. J Cardiothorac Vasc Anesth. 2016 Oct;30(5):1228-33. doi: 10.1053/j.jvca.2016.06.007. Epub 2016 Jun 8. PMID 27640893
- [Result] Afzal MR, Okabe T, Koppert T, Tyler J, Houmsse M, Augostini RS, Hummel JD, Kalbfleisch SJ, Iyer MH, Flores AS, Bhandary S, Dimitrova G, Elsayed-Awad H, Fiorini K, Gorelik L, Perez W, Saklayen S, Stein E, Turner K, Franklin NP, Ryu JN, Bhatt A, Weiss R, Daoud EG, Essandoh M. Implantation of subcutaneous defibrillator is feasible and safe with monitored anesthesia care. Pacing Clin Electrophysiol. 2019 Dec;42(12):1552-1557. doi: 10.1111/pace.13838. Epub 2019 Nov 18. PMID 31702059
- [Result] Ziacchi M, Bisignani G, Palmisano P, Scalone A, Martignani C, Elvira Mocavero P, Caravati F, Della Cioppa N, Mazzuero A, Pecora D, Vicentini A, Landolina ME, Debonis S, Scimia P, Lovecchio M, Valsecchi S, Diemberger I, Droghetti A. Serratus anterior plane block in subcutaneous implantable cardioverter defibrillator implantation: A case-control analysis. J Cardiovasc Electrophysiol. 2020 Jan;31(1):144-149. doi: 10.1111/jce.14293. Epub 2019 Dec 3. PMID 31778266
- [Result] Miller MA, Garg J, Salter B, Brouwer TF, Mittnacht AJ, Montgomery ML, Honikman R, Arkonac DE, Choudry S, Dukkipati SR, Reddy VY, Weiner MM. Feasibility of subcutaneous implantable cardioverter-defibrillator implantation with opioid sparing truncal plane blocks and deep sedation. J Cardiovasc Electrophysiol. 2019 Jan;30(1):141-148. doi: 10.1111/jce.13750. Epub 2018 Oct 22. PMID 30230098
- [Result] Uran C, Giojelli A, Borgogna DA, Morello G, Marullo F, Iodice P, Greco A, Accogli M, Guido A, Palmisano P. Ultrasound-guided serratus anterior plane block combined with parasternal block in subcutaneous implantable cardioverter defibrillator implantation: Results of a pilot study. Pacing Clin Electrophysiol. 2020 Jul;43(7):705-712. doi: 10.1111/pace.13944. Epub 2020 Jun 3. PMID 32420626